CLINICAL TRIAL: NCT01522066
Title: Comparison of the Effectiveness of Single-shot Local Anesthetic Delivery Versus Double-shot Local Anesthetic Delivery Via a Perineural Catheter
Brief Title: Catheter-over Needle: Outpatient Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at institution
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro000027421
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Local Anesthesia; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perineural catheter (Experimental): Local anesthetic will be delivered through an indwelling perineural catheter
  Interventions: Procedure: Perineural catheter
- Single-shot block (Active Comparator): Local anesthetic will be delivered by the conventional, single-shot method.
  Interventions: Procedure: Single-shot block

INTERVENTIONS:
Procedure: Perineural catheter — Patients in the experimental group will receive a single dose of local anesthetic though an indwelling catheter both before and after surgery.
  Arms: Perineural catheter
Procedure: Single-shot block — Patients in the control group will receive a single shot of local anesthetic, in standard fashion, before surgery.
  Arms: Single-shot block

SUMMARY:
An alternative to general anesthesia - which puts a patient completely to sleep - is regional anesthesia, where local anesthetic is injected under the skin to freeze or 'block' a nerve or set of nerves. This method allows a patient to be awake during surgery and avoids any unpleasant after-effects of general anesthetic. A regional block is normally performed by inserting a needle under the skin so that the needle tip is near the nerve to be blocked, followed by injection of a single shot of enough local anesthetic to block any sensation that the nerve normally provides. Although regional nerve blocks provide pain relief during a surgical procedure, they eventually wear off, occasionally leaving the patient to contend with localized pain in the part of the body that was operated on. In these cases, over-the-counter painkillers like Tylenol or Advil may not be strong enough to completely take away the pain. We believe that, instead of giving a single shot of anesthetic, patients can be fitted with a catheter - a thin, flexible tube - that can be used to deliver one dose of local anesthetic to block the nerve before surgery and which could also be used to deliver a second dose of anesthetic just prior to discharge from the hospital. This way, the patient still only receives one needle poke, but their pain can be better managed following surgery. Our study will compare the post-nerve block pain profiles of individuals who have received a single-shot injection of local anesthetic versus those who have received two doses via the catheter delivery method.

DETAILED DESCRIPTION:
Background: Local anesthetic (LA) may be delivered by a single injection or by continuous infusion through an indwelling catheter. A downside of the single-shot technique is that the LA has a limited duration of action, meaning that, after discharge, patients sometimes have to contend with post-surgical pain that limits their activities and reduces their quality of life. Occasionally, a supplementary dose of analgesic, such as morphine or a LA, will be administered, either intravenously or via single injection. We speculate that, rather than using a single injection, post-operative pain management may be better controlled by installing a perineural catheter pre- or intra-operatively, which would allow a flexible schedule of LA delivery post-operatively and enable clinicians to tailor an analgesia regimen to the patient's needs. Our aim is to compare the effectiveness of a double-shot anesthetic infusion - one to block the nerve and another to provide postoperative analgesia - to the conventional single-shot method in controlling pain following a regional nerve block.

Study objective: To assess the value of a catheter-delivered supplementary infusion of LA to control postoperative pain after a regional block.

Hypothesis: Patients who have received a regional nerve block will experience less post-surgical pain when a second shot of LA is delivered through a perineural indwelling catheter just prior to discharge.

Study procedures: We will recruit patients who are scheduled to undergo surgery that requires a regional block of the upper extremity. We anticipate recruiting thirty individuals; the control group will receive one dose of LA using the conventional single-shot method, and the study group will be fitted with a perineural catheter through which one dose of LA will be delivered prior to surgery and another just before discharge from the hospital.

On the day of surgery, participating patients will be taken to the regional block area. Control group patients will be given a single injection of LA, under ultrasound guidance, to block the appropriate target nerve(s). These patients will undergo surgery and post-anesthesia recovery as per standard procedures. For patients in the experimental group, the attending anesthesiologist will, under ultrasound guidance, insert a perineural catheter at an appropriate location to block the target nerve. Once the catheter is in place, a single dose of LA will be delivered to block the target nerve, and the catheter will remain in the patient throughout the procedure. In the post-anesthesia recovery area, patients with a catheter will receive a second bolus infusion of the same LA. When the patient is approved for discharge, the catheter will be removed, the insertion site cleaned, and the patient will be allowed to go home.

A research assistant ask patients to rate their pain using a 0-10 numerical rating scale: 1) prior to delivery of the first dose of LA, 2) immediately following surgery (just before the second anesthetic infusion for experimental group patients), and 3) immediately before discharge from the hospital (after the second anesthetic infusion for experimental group patients). On the day after surgery, the research assistant will contact patients in both groups and will ask them to rate their pain over the 24-hour post-operative period. Pain reporting at these four time points will provide us with a comprehensive assessment of patient comfort after their regional nerve block and whether the second infusion of LA was effective at alleviating post-operative pain.

Primary outcomes:

1. Postoperative pain levels
2. Patient comfort at home

Inclusion criteria: Adult; scheduled for surgery that requires peripheral nerve blockade.

Exclusion criteria: Failure to provide informed consent; allergy to LA; neurological pathology and/or deficit in the block region.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 yrs)
* Scheduled for surgery that requires peripheral nerve blockade

Exclusion Criteria:

* Failure to provide informed consent
* Allergy to local anesthetic
* Neurological pathology and/or deficit in the block region

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain levels | 24 hours following surgery
  Pain levels at surgery site following surgery (up to 24 hours post-surgery) will be assessed.

SECONDARY OUTCOMES:
Patient comfort at home | Post-operative period (approx. 24 hrs following surgery)
  Patient pain levels and effects on daily living/activities will be assessed following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Tsui, MD, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Ip VH, Tsui BC. The catheter-over-needle assembly facilitates delivery of a second local anesthetic bolus to prolong supraclavicular brachial plexus block without time-consuming catheterization steps: a randomized controlled study. Can J Anaesth. 2013 Jul;60(7):692-9. doi: 10.1007/s12630-013-9951-5. Epub 2013 May 1. PMID 23637033